CLINICAL TRIAL: NCT05110677
Title: Pilot Study of Topographic Imaging of the Gastrocnemius Muscle in Patients With PAD Using Non-invasive Multispectral Optoacoustic Tomography (MSOT) as a 3D Reconstruction Based on Longitudinal 2D Measurements
Brief Title: Pilot Study of Topographic Imaging of the Calf Muscle in Patients With PAD Using 3D Reconstruction of MSOT Images
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Erlangen (Other)
Collaborators: Department of Pediatrics and Adolescent Medicine, University Hospital Erlangen, Erlangen, Germany (Unknown); Division of Computer Assisted Medical Interventions, German Cancer Research Center, Heidelberg, Germany (Unknown)
Responsible Party: Principal Investigator, Ulrich Rother, PD Dr. med., University Hospital Erlangen
Other Study IDs: MSOT_PAD_3D
Record Dates: First submitted 2021-10-12; First posted 2021-11-08 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Peripheral Vascular Diseases; Peripheral Arterial Disease
Keywords: Peripheral Vascular Disease; Peripheral Arterial Disease; Multispectral Optoacoustic Tomography; MSOT; PAD; Claudicatio intermittens; Critical Limb Ischemia; CLI; Diagnostic imaging; Color-Coded Duplex Sonography; CCDS; Non-invasive diagnostic procedure; non-invasive diagnostic; noninvasive diagnostic; 3D imaging; three-dimensional imaging; three-dimensional diagnostic; 3D diagnostic; tattoo tomography; optical pattern
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Multispectral Optoacoustic Tomography (MSOT) and B-Mode Ultrasound of the Musculus gastrocnemius of the affected leg in PAD patients or one leg in healthy volunteers (total 1 site)
  Physical assessment: Color-Coded Duplex Sonography/treadmill examination to determine actual walking distance/Ankle-Brachial-Index/defined walking distance of 150 meters under medical supervision
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography (MSOT) — non-invasive transcutaneous imaging of subcellular muscle components

SUMMARY:
The aim of this explorative pilot study is to present muscle perfusion of the lower extremity in patients with PAD using the Multispectral Optoacoustic Tomography (MSOT) method to build a 3D reconstruction of the calf muscle. This study aims to show the feasibility of 3D reconstruction of this non-invasive method. Advantages in diagnostics for patients with PAD and three-dimensional tomography representation of the perfusion situation based on muscle oxygenation will be evaluated.

DETAILED DESCRIPTION:
Functional imaging diagnostics is becoming increasingly important due to the steadily growing knowledge of physiological processes in many diseases. Also in peripheral arterial occlusive disease (PAD), new insights into the pathomechanism of the disease are continuously being gained. This also increases the need for new non-invasive imaging methods that are able to visualize the functional level of the disease progression and thus make it possible to diagnose it at an early stage.

Recent studies indicate that it may be feasible to use multispectral optoacoustic tomography (MSOT) to visualize hemodynamics as well as the fibrotic muscle remodeling process in PAD. For a better understanding of the distribution pattern , the exploration of a 3D technique is a next necessary step in imaging. This may show a possible existing heterogeneity of these molecules.

Holzwarth et al. were already able to gain knowledge about the 3D reconstruction from 2D photoacoustic image slices using an optical pattern and the method's feasibility using phantoms as well as in-vivo measurements of the forearm in healthy volunteers.

The aim of this exploratory pilot project is to bring these previous findings together and to image muscle perfusion of the lower extremity in three dimensions using the MSOT method and to verify its feasibility. The advantage of 3D imaging is, beyond the anatomical topography of the muscle, to map a three-dimensional representation of the perfusion situation based on muscle oxygenation.

For this purpose, six patients of different symptomatic PAD stages and a healthy control of two volunteers will be included and examined by means of longitudinal MSOT scans in the area of the gastrocnemius muscle. To evaluate the current stage of the disease or to exclude relevant PAD in the healthy control population, non-invasive examination measures commonly used in routine diagnostics of PAD will be applied. In addition to the relevant risk factors/adjacent diseases and the current medication intake, these include the recording of the ankle-brachial index (ABI), color-coded duplex sonographic vascular imaging (CCDS) and a treadmill examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with manifest PAD stages II-IV according to Fontaine or healthy volunteers
* Adult (>18 years) persons who are able to give their consent

Exclusion Criteria:

* Patients with PAD stage I according to Fontaine
* Healthy volunteers with pre-existing diabetes mellitus, chronic renal failure, or abnormal ABI
* Underage persons
* Missing consent form
* Exclusion due to safety concerns of the study physician (patient with a physical, mental or psychiatric illness which, in the opinion of the study physician, would compromise the safety of the patient or the quality of the data and thus make the patient an unsuitable candidate for the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with PAD IIa/IIb/III/IV according to Fontaine who come in for a routine presentation of the the vascular surgery consultation hours.
  Healthy volunteers with
  * no PAD previously known
  * no diabetes mellitus previously known
  * no chronic renal insufficiency previously known
  * no symptoms in the sense of a Claudicatio intermittens
  * ABI with normal value who are recruited by clinic notices.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
MSOT topogram showing MSOT parameters from 660 up to 1100 nm of the gastrocnemius muscle | single time point (1 day)
  MSOT topogram using 3D reconstruction based on longitudinal 2D scans trough an optical pattern showing MSOT parameters from 660 up to 1100 nm of the gastrocnemius muscle

SECONDARY OUTCOMES:
Acquisition of the quantitative hemoglobin signal (oxygenated/deoxygenated) | single time point (1 day)
  This Outcome is measured non-invasively by MSOT, the single wavelengths are spectrally unmixed
Acquisition of the quantitative fibrosis signals (collagen/lipid) | single time point (1 day)
  This Outcome is measured non-invasively by MSOT, the single wavelengths are spectrally unmixed
3D reconstruction of the longitudinal measurements using two different pattern designs | single time point (1 day)
  This Outcome is measured non-invasively by MSOT. A foil imprinted with an "N" is applied and fixed over the calf muscle. Three longitudinal 2D measurements are made or repeated until a promising result is obtained. The same procedure is repeated with a foil imprinted with a trident.
Acquisition of static 2D MSOT measurements before and after gait exposure | single time point (1 day)
  This Outcome is measured non-invasively by MSOT. An initial measurement is taken at rest. Subsequently, the patient will complete a defined walking distance of 150 meters under medical supervision. Afterwards, the medial head of the gastrocnemius muscle is measured again.
Validation of the accuracy of the MSOT 3D reconstruction using an overlay from MRA | single time point (1 day)
  This Outcome is only realized in participants who received an magnetic resonance angiography regardless of study participation
Acquisition of the flow profile of the common femoral artery and popliteal artery using CCDS | single time point (1 day)
  This Outcome is measured non-invasively by standardized vascular sonography
Acquisition of the Ankle-Brachial-Index | single time point (1 day)
  This Outcome is measured non-invasively by standardized clinical assessment according to the according to the recommendation from the S3 guideline for PAD of the German Association for Angiology ("Deutsche Gesellschaft für Angiologie") dated November 30, 2015
Acquisition of the current walking distance standardized by treadmill examination | single time point (1 day)
  This Outcome is measured by a standardized treadmill examination (excluding PAD patients in chronic critical stage III or IV according to Fontaine) ideally with 3km/h and 12% incline
Acquisition of the PAD stage according to Fontaine and Rutherford | single time point (1 day)
  This Outcome is acquired by actual recommendation from national and international guidelines
Recording of relevant patient data from the patient's file | single time point (1 day)
  Preexisting disorders, previous performed operations on vessels, current medication, radiological TransAtlantic InterSociety Consensus classification

CONTACTS AND LOCATIONS:
Locations (1):
- University of Erlangen, Vascular Surgery, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Signorelli SS, Vanella L, Abraham NG, Scuto S, Marino E, Rocic P. Pathophysiology of chronic peripheral ischemia: new perspectives. Ther Adv Chronic Dis. 2020 Feb 5;11:2040622319894466. doi: 10.1177/2040622319894466. eCollection 2020. PMID 32076496
- [Background] Karlas A, Kallmayer M, Fasoula NA, Liapis E, Bariotakis M, Kronke M, Anastasopoulou M, Reber J, Eckstein HH, Ntziachristos V. Multispectral optoacoustic tomography of muscle perfusion and oxygenation under arterial and venous occlusion: A human pilot study. J Biophotonics. 2020 Jun;13(6):e201960169. doi: 10.1002/jbio.201960169. Epub 2020 Mar 25. PMID 32134550
- [Background] Holzwarth N, Schellenberg M, Grohl J, Dreher K, Nolke JH, Seitel A, Tizabi MD, Muller-Stich BP, Maier-Hein L. Tattoo tomography: Freehand 3D photoacoustic image reconstruction with an optical pattern. Int J Comput Assist Radiol Surg. 2021 Jul;16(7):1101-1110. doi: 10.1007/s11548-021-02399-w. Epub 2021 May 16. PMID 33993409

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT05110677/Prot_SAP_000.pdf